CLINICAL TRIAL: NCT00729547
Title: The Therapeutic Efficacy of Frontal EEG Asymmetry Neurofeedback in Depression
Brief Title: The Therapeutic Efficacy of Neurofeedback in Depression
Acronym: neurofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: Korea Research Foundation (Other); Kyunghee University (Other)
Responsible Party: Hyun Taek Kim/Professor, Department of Psychology, Korea University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KRF-2005-079-HS0012
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2006-09

CONDITIONS: Depression
Keywords: Depression; Biofeedback; Psychophysiology
MeSH Terms: conditions — Depression | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Psychotherapy placebo session
  Interventions: Behavioral: Psychotherapy placebo
- 1 (Experimental): Neurofeedback training which enhance left frontal alpha wave.
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — enhance relative activity level of left frontal activity
  Other Names: Asymmetry training
  Arms: 1
Behavioral: Psychotherapy placebo — These sessions consisted of additional assessment, interpretation of the test results and providing information on course and treatment of mood disorder.
  Arms: 2

SUMMARY:
The investigators examined the therapeutic efficacy of neurofeedback in depression subjects. The investigators hypothesize that 5 weeks neurofeedback training will be able to alleviate depressive symptoms.

DETAILED DESCRIPTION:
Subject

* Fulfilled DSM-IV criteria for depressive disorders.
* Persons who had organic disorders were excluded.
* Who had been treated by psychoactive drugs for at least 2 months prior to the study were excluded.

Design

* Subjects were randomly assigned to two groups (EEG biofeedback /psychotherapy placebo) by block randomization.
* EEG biofeedback training was provided for 5 weeks(10 sessions, twice per week). Each training session was composed of 6 four minute trials followed by 5 thirty second rest periods
* Psychotherapy placebo session was provided for 5 weeks. These sessions consisted of additional assessment, interpretation of the test results and providing information on course and treatment of mood disorder.
* After subjects completed the training, they participated in a month-long (twice per week) self-training session to maintain a similar mental state during neurofeedback training sessions without feedback system's assistance.
* Subjects who had finished the psychotherapy placebo were referred to other therapists as necessary.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of mood disorder
* right handed
* current BDI-2 score exceed 10

Exclusion Criteria:

* with psychotic symptom
* with organic disorders
* treated by psychoactive drugs for at least 2 months prior to the study
* history of pathologic alcohol use

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
frontal EEG asymmetry indexes | 5 weeks

SECONDARY OUTCOMES:
BDI-2 | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyuntaek Kim, PHD, Principal Investigator — Department of Psychology, Korea university
Locations (1):
- Department of Oriental Neuropsychiatry, Kyunghee Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Hammond DC. Neurofeedback with anxiety and affective disorders. Child Adolesc Psychiatr Clin N Am. 2005 Jan;14(1):105-23, vii. doi: 10.1016/j.chc.2004.07.008. PMID 15564054
- [Background] Rosenfeld JP. An EEG biofeedback protocol for affective disorders. Clin Electroencephalogr. 2000 Jan;31(1):7-12. doi: 10.1177/155005940003100106. No abstract available. PMID 10638347
- [Result] Kumano H, Horie H, Shidara T, Kuboki T, Suematsu H, Yasushi M. Treatment of a depressive disorder patient with EEG-driven photic stimulation. Biofeedback Self Regul. 1996 Dec;21(4):323-34. doi: 10.1007/BF02214432. PMID 9031711
- [Result] Rosenfeld JP, Cha G, Blair T, Gotlib IH. Operant (biofeedback) control of left-right frontal alpha power differences: potential neurotherapy for affective disorders. Biofeedback Self Regul. 1995 Sep;20(3):241-58. doi: 10.1007/BF01474516. PMID 7495918
- [Result] Saxby E, Peniston EG. Alpha-theta brainwave neurofeedback training: an effective treatment for male and female alcoholics with depressive symptoms. J Clin Psychol. 1995 Sep;51(5):685-93. doi: 10.1002/1097-4679(199509)51:53.0.co;2-k. PMID 8801245
- See also: click here to review subject recruiting and information on this study — http://www.psychonews.co.kr
- See also: click here to see brief description of the department of psychology at Korea university — http://psy.korea.ac.kr
- See also: click here to review the location of this study and the policy of IRB — http://www.khmc.or.kr